CLINICAL TRIAL: NCT06971159
Title: Clinical, Metabolic, Physical, Functional, Biochemical, and Cardiovascular Evaluation in Individuals With Obesity After Performing Systemic Vibratory Therapy and Osteopathic Manipulative Treatment
Brief Title: Systemic Vibratory Therapy and Osteopathic Manipulative Treatment in Individuals With Obesity
Acronym: SVT and OMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratorio de Vibraçoes Mecanicas e Praticas Integrativas (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Universidade do Estado do Rio de Janeiro - UERJ (Unknown); Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 30649620.1.0000.5259
Record Dates: First submitted 2025-04-28; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Obesity
Keywords: systemic vibratory therapy; osteopathic manipulative treatment; obesity
MeSH Terms: conditions — Obesity | interventions — Manipulation, Osteopathic; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Systemic Vibratory Therapy Group (Experimental): The SVT interventions occur on the alternating vibrating platform (VP) (Novaplate fitness evolution, DAF Produtos Hospitalares Ltda, São Paulo). The individual is positioned barefoot, with 130º of knee flexion, frequency of 30 Hz, peak-to-peak displacement of 2.5 mm. The individuals will perform 9 sets of SVT consisting of 1 minute of vibration with 1 minute of rest, totaling 17 minutes of exercise.
  Interventions: Device: Systemic vibratory therapy
- Osteopathic manipulative treatment group (Experimental): Osteopathic manipulative treatment consists of the following techniques: i) suboccipital inhibition technique (5 minutes) and suboccipital decompression (3 minutes); ii) myofascial release technique of the cervical spinal muscles (2 minutes); iii) diaphragm muscle release technique (5 minutes), totaling 15 minutes of treatment.
  Interventions: Other: Osteopathic manipulative treatment
- Systemic vibratory therapy combined with osteopathic manipulative treatment (Experimental): In this group, individuals undergo a combined treatment. First, systemic vibration therapy is performed (according to the protocol mentioned in the systemic vibration therapy group) and then osteopathic manipulative treatment is performed (according to the protocol mentioned in the osteopathic manipulative treatment group).
  Interventions: Device: Systemic vibratory therapy; Other: Osteopathic manipulative treatment
- Osteopathic manipulative treatment combined with systemic vibratory therapy (Experimental): In this group, individuals undergo a combined treatment. First, osteopathic manipulative treatment is performed (according to the protocol mentioned in the osteopathic manipulative treatment group) and then systemic vibration therapy is performed (according to the protocol mentioned in the systemic vibration therapy group).
  Interventions: Device: Systemic vibratory therapy; Other: Osteopathic manipulative treatment
- Sham group (Sham Comparator): In the sham group, simulation of the SVT is performed, where the individual is stand on the PV, barefoot, with 130º of knee flexion and remain in this position during the active periods of the protocol, with the PV turned off, emitting only a vibration simulation through a device attached to it and the OMT in which the researcher will perform a treatment simulation by simply placing his hands on the suboccipital, cervical and diaphragm muscle regions, without exercising any therapeutic intention.
  Interventions: Other: Sham

INTERVENTIONS:
Device: Systemic vibratory therapy — Systemic vibratory therapy is an intervention in which mechanical vibration, generated by the vibrating platform, is transmitted to the whole-body of the individual generating whole-body vibration exercise.
  Arms: Osteopathic manipulative treatment combined with systemic vibratory therapy; Systemic Vibratory Therapy Group; Systemic vibratory therapy combined with osteopathic manipulative treatment
Other: Osteopathic manipulative treatment — Osteopathic manipulative treatment is defined by the WHO as a diagnostic and therapeutic method that uses manual contact for these purposes. It concerns the relationship between body, mind and spirit in health and illness, emphasizing the structural and functional integrity of the body and the body's intrinsic tendency to direct itself towards healing.
  Arms: Osteopathic manipulative treatment combined with systemic vibratory therapy; Osteopathic manipulative treatment group; Systemic vibratory therapy combined with osteopathic manipulative treatment
Other: Sham — In the sham group, the interventions are simulated, as described in the sham group protocol.
  Arms: Sham group

SUMMARY:
Studies have demonstrated a strong relationship between physical inactivity and the presence of obesity and other cardiovascular risk factors such as hypertension, insulin resistance, diabetes, dyslipidemia, and metabolic syndrome. On the other hand, regular physical exercise has been recommended for the prevention and treatment of cardiovascular diseases, their risk factors, and other chronic conditions.

Systemic vibratory therapy (SVT) and osteopathic manipulative treatment (OMT) has been proposed as alternative therapies for this population.

The aim of this project is to assess clinical, metabolic, physical, functional and cardiovascular parameters, in individuals with obesity undergoing systemic vibratory therapy and the osteopathic manipulative treatment.

The clinical evaluation included measurements of heart rate variability, systemic blood pressure, heart rate, respiratory rate, oxygen saturation, handgrip dynamometry, the BORG scale, NPS (Numerical Pain Scale), and RPE (Rating of Perceived Exertion) scale; anthropometric measurements including neck, abdominal, hip, arm, thigh and calf circumferences; as well as body composition assessment and anterior trunk flexibility. Additional information was collected, including age, sex, smoking status, physical inactivity, associated comorbidities and medication use.

Laboratory analyses included a complete blood count, total cholesterol and its fractions, triglycerides, creatinine, uric acid, cortisol, glucose, insulin, growth hormone, vitamin D, and other relevant blood parameters. Questionnaires were administered to access the level of physical activity.

Participants were randomized into five groups: systemic vibratory therapy group (SVT), osteopathic manipulative treatment group (OMT), SVT+OMT, OMT+SVT, and control group. The parameters mentioned above are collected before the intervention (baseline), immediately after one session of the respective intervention (acute effect), and after 12 sessions (cumulative effect).

DETAILED DESCRIPTION:
For anamnesis, data is collected from participants, including age, sex, smoking status, alcohol consumption, presence and type of diabetes mellitus, presence of systemic arterial hypertension, associated comorbidities, medication use, history of COVID-19, and physical inactivity.

Clinical assessments are conducted before and after the 12 sessions of systemic vibratory therapy, including measurements of systemic blood pressure, heart rate variability, heart rate, oxygen saturation, respiratory rate, the BORG scale and the Numeric Pain Scale (NPS). Anthropometric measurements were collected, including neck, arm, abdominal, hip, thigh and ankle circumferences, as well as body composition distribution assessed via bioelectrical impedance, and lumbar spine flexibility via anterior trunk flexion test.

Laboratory analyses of relevant biomarkers, the HOMA-IR index, and anthropometric indicators were also evaluated. Questionnaires were administered to assess quality of life.

Neuromuscular activity is assessed using handgrip strength via a manual dynamometer.

Heart rate variability is assessed using a heart rate monitor.

Patients were positioned on the platform base under the supervision of a healthcare professional to perform the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes;
* Individuals with obesity;
* Over 18 years old.

Exclusion Criteria:

* Body mass index (BMI) < 30 kg/m2;
* Uncontrolled untreated hypertension, with elevated systemic blood pressure levels (≥180 x 110 mmHg);
* Cardiovascular diseases (myocardial infarction/stroke), in the last 6 months;
* Atrial fibrillation;
* History of spine surgery;
* Neurological, rheumatological diseases or osteoarticular lesions that hinder movements of the vibrating platform (VP);
* Serious or disabling diseases, at the discretion of the investigator;
* Individuals who refuse to sign the Informed Consent Form (ICF) to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2030-05-30 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | Heart rate variability analyzed at the baseline (day 1), immediately after the intervention (day 1), and after 12 sessions of the intervention (day 12).
  Heart rate variability indices analyzed using a heart rate monitor. Indices are analyzed in the time domain (mean RR, SDNN, mean HR, RMSSD, pNN50), frequency domain (LF, HF, LF/HF ratio), and non-linear methods (SD1, SD2, SD2/SD1 ratio).
Heart rate | From enrollment to the end of treatment at 6 weeks.
  Heart rate (unit of measurement in beats per minute) is measured using the G-tech Led Digital Finger Oximeter. Resting, training, and recovery heart rates: These will be investigated to assess the intensity of physical effort in terms of the percentage of training achieved.
Systemic arterial pressure | From enrollment to the end of treatment at 6 weeks.
  Systemic arterial pressure (unit of measurement in mmHg) is measured with the individual seated, after 5 minutes of rest, with an automatic blood pressure monitor by OMRON, model HEM7113 (Japan), positioned on the individual's left arm, which should be relaxed and at heart level. The cuff will be positioned 3 to 4 cm above the antecubital fossa, with the elbow slightly flexed and the forearm in supination. This measurement will occur 3 times, with a 1-minute interval between them. The average of the three measurements will be considered for analysis.
Anthropometric measurements | Analyzed at the baseline (day 1) and after 12 sessions of the intervention (day 12).
  Anthropometric measurements, as circumferences were assessed to evaluate the distribution of fat and other physical characteristics. The circumference measurements will be taken at the following sites, measured in centimeters (cm): neck, abdominal, hip, arm, thigh and calf circumferences.
Body Mass Index (BMI) | From enrollment to the end of treatment at 6 weeks.
  Body Mass Index (BMI) is a clinical index that is used in bioimpedance to assess a person's weight. BMI is calculated by dividing the weight (in kg) by the height (in meters) squared. Unit of measure: kilograms per square meter (kg/m²).
Waist-to-Hip Ratio (WHR) | From enrollment to the end of treatment at 6 weeks.
  The ratio of the circumference of the waist to the circumference of the hips, used as an indicator of cardiovascular risk. WHR was calculated by dividing the waist circumference in centimeters by the hip circumference. It is an element for the prognosis of cardiovascular events in adults. The cut-off index for cardiovascular risk is less than 0.85 for women and 0.90 for men. The unit of measurement is unitless.
Waist-to-Height Ratio (WHtR) | From enrollment to the end of treatment at 6 weeks.
  The ratio of the circumference of the waist to height, used as an indicator of metabolic and cardiovascular risk. Height was measured using a vertical stadiometer graduated in centimeters and millimeters. Waist circumference was assessed using a tape measure graduated in centimeters and millimeters. The tape measure was placed midway between the iliac crest and the last rib. This anatomical point has the strongest correlation with abdominal adiposity. The values obtained were stratified into three categories: between 0.40 and 0.44 (lowest % fat, below the risk threshold); between 0.45 and 0.50 (moderate risk); between 0.50 and 0.56 (above the risk threshold). The unit of measurement is unitless.
Conicity Index | From enrollment to the end of treatment at 6 weeks.
  Conicity index is a measure of body fat distribution, particularly visceral fat, calculated using body circumference measurements. The C Index (CI) was determined based on the measurement of body mass, height and waist circumference, in meters, representing an indicator of abdominal obesity, and is based on the principle that some people accumulate fat around the abdomen, with the consequent change in body shape. This index is calculated using the formula: C Index = waist circumference (m)/(0.109 x (√ body mass (kg)/height (m))). For the classification of cardiovascular risk, values ≥ 1.18 for women and ≥ 1.25 for men are determined. The unit of measurement is unitless.
Basal Metabolic Rate | From enrollment to the end of treatment at 6 weeks.
  Basal Metabolic Rate will be analyzed using a Tetrapolar Bioelectrical Impedance Analyzer (InBody 370, BIOSPACE, Republic of Korea). The analyzer performs impedance measurements across five body segments (right arm, left arm, trunk, right leg, and left leg) using three different frequencies (5, 50, and 500 kHz), and provides separate body mass readings for each segment. The device provides separate body mass readings for different body segments, being able to estimate the basal metabolic rate. The basal metabolic rate is directly proportional to the weight and amount of muscle. It was calculated from predictive formulas using the results of the body composition, and involves the data of age, sex and physical activity that is entered into the scale. Unit of measure: kilocalories per day (kcal/day).
Visceral Fat Area | From enrollment to the end of treatment at 6 weeks.
  The visceral fat area of the body composition will be analyzed using a Tetrapolar Bioelectrical Impedance Analyzer (InBody 370, BIOSPACE, Republic of Korea). The analyzer performs impedance measurements across five body segments (right arm, left arm, trunk, right leg, and left leg) using three different frequencies (5, 50, and 500 kHz), and provides separate body mass readings for each segment. Unit of measure: square centimeters (cm²).
Body Fat Percentage | From enrollment to the end of treatment at 6 weeks.
  The Body fat percentage of the body composition will be analyzed using a Tetrapolar Bioelectrical Impedance Analyzer (InBody 370, BIOSPACE, Republic of Korea). The analyzer performs impedance measurements across five body segments (right arm, left arm, trunk, right leg, and left leg) using three different frequencies (5, 50, and 500 kHz), and provides separate body mass readings for each segment. Unit of measure: Expressed as a percentage (%).
Lean Body Mass, Fat Mass, and Skeletal Muscle Mass | From enrollment to the end of treatment at 6 weeks.
  The measures of body composition will be analyzed using a Tetrapolar Bioelectrical Impedance Analyzer (InBody 370, BIOSPACE, Republic of Korea). The analyzer performs impedance measurements across five body segments (right arm, left arm, trunk, right leg, and left leg) using three different frequencies (5, 50, and 500 kHz), and provides separate body mass readings for each segment. The following body composition components will be measured: Lean Body Mass: Measured in kilograms (kg). Fat Mass: Measured in kilograms (kg). Skeletal Muscle Mass: Measured in kilograms (kg).
Total Body Water | From enrollment to the end of treatment at 6 weeks.
  The measure of the Total Body Water of the body composition will be analyzed using a Tetrapolar Bioelectrical Impedance Analyzer (InBody 370, BIOSPACE, Republic of Korea). The analyzer performs impedance measurements across five body segments (right arm, left arm, trunk, right leg, and left leg) using three different frequencies (5, 50, and 500 kHz), and provides separate body mass readings for each segment. Unit of Measured: in liters (L).
Oxygen saturation | From enrollment to the end of treatment at 6 weeks.
  Oxygen saturation (unit of measurement in percentage) is measured using the G-tech Led Digital Finger Oximeter, with the individual seated, after 5 minutes of rest. This measurement will occur 3 times, with a 1-minute interval between them. The average of the three measurements will be considered for analysis.
Respiratory rate | From enrollment to the end of treatment at 6 weeks.
  Respiratory rate (unit of measurement in cycles per minute) is measured by observing how many respiratory cycles are performed per minute, with the individual in a lying, sitting and standing position.

SECONDARY OUTCOMES:
Funcional parameters | Analyzed at the baseline (day 1) and after 12 sessions of the intervention (day 12).
  Timed Up and Go test - The volunteer sits on a chair, is ordered to stand up and walk to a mark on the floor (distance of 3 meters), turns and returns to the chair, sits on the chair, the time spent is measured in seconds and thousandths of a second with a stopwatch.
Metabolic Biomarkers | From enrollment to the end of treatment at 6 weeks.
  Peripheral blood samples were aseptically collected using an intravenous catheter inserted into an antecubital vein. The blood was separated by centrifugation. Serum cortisol levels were assessed in serum samples using standard laboratory techniques after an 8-hour fasting period. Unit of Measure: µg/dL. Sample collection was conducted at the Clinical Analysis Laboratory (Cápsula) of PPC-UERJ, always during the same shift, no later than 8:00 AM.
Hormonal Biomarkers | From enrollment to the end of treatment at 6 weeks.
  Peripheral blood samples were aseptically collected using an intravenous catheter inserted into an antecubital vein. The blood was separated by centrifugation. Insulin, and growth hormone (HGH) levels were assessed in serum samples using standard laboratory techniques after an 8-hour fasting period. Unit of Measure: ng/mL. Sample collection was conducted at the Clinical Analysis Laboratory (Cápsula) of PPC-UERJ, always during the same shift, no later than 8:00 AM.
Uric Acid Levels | From enrollment to the end of treatment at 6 weeks.
  Peripheral blood samples were aseptically collected using an intravenous catheter inserted into an antecubital vein. The blood was separated by centrifugation. Serum uric acid levels were measured in serum samples collected after an 8-hour fasting period. Unit of Measure: mg/dL. Sample collection was conducted at the Clinical Analysis Laboratory (Cápsula) of PPC-UERJ, always during the same shift, no later than 8:00 AM.
Lipid Profile and Fasting Blood Glucose | From enrollment to the end of treatment at 6 weeks.
  Peripheral blood samples were aseptically collected using an intravenous catheter inserted into an antecubital vein. The blood was separated by centrifugation. Total cholesterol, low-density lipoprotein (LDL), high-density lipoprotein (HDL), and triglyceride levels were measured in serum samples, and fasting blood glucose levels were measured in plasma samples. All measures collected after an 8-hour fasting period. Unit of Measure: mg/dL Sample collection was conducted at the Clinical Analysis Laboratory (Cápsula) of PPC-UERJ, always during the same shift, no later than 8:00 AM.
Glycated Hemoglobin (HbA1c) | From enrollment to the end of treatment at 6 weeks.
  Peripheral blood samples were aseptically collected using an intravenous catheter inserted into an antecubital vein. The blood was separated by centrifugation. Glycated hemoglobin (HbA1c, %) levels were measured in plasma samples collected after an 8-hour fasting period. Unit of Measure: % (for HbA1c). Sample collection was conducted at the Clinical Analysis Laboratory (Cápsula) of PPC-UERJ, always during the same shift, no later than 8:00 AM.
Muscle strength | From enrollment to the end of treatment at 6 weeks.
  The Lafayette dynamometer (hand grip dynamometers model j00105) will be used. Participants will be seated with their feet on the floor, their arm in adduction and elbow flexed at 90°, their forearm in a neutral position and their wrist extended between 0° and 30°. Three repetitions of maximum grip of 3 seconds will be performed, with a recovery period of 60 seconds between repetitions.
Pain Level | From enrollment to the end of treatment at 6 weeks.
  It is essential to know the participant's pain, and to assess pain, scales such as the visual analogue scale (VAS) will be used, which consists of a ruler divided into eleven equal parts from zero to ten, where the individual is expected to make the equivalence according to the level of their pain through the numerical classification (zero corresponding to the least and ten to the greatest pain).
Physical activity | From enrollment to the end of treatment at 6 weeks.
  Assessing the level of physical activity is essential to assess an individual's current health conditions and helps to determine which exercises can be part of their routine. This assessment allows the identification of physical and biological limitations, in addition to finding signs of some diseases. Thus, to classify the level of physical activity of the individual, duly validated questionnaires will be used, such as the International Physical Activity Questionnaire (IPAQ), which allows the estimation of the weekly time spent in moderate and vigorous physical activities in different contexts of daily life. The short version will be applied, consisting of 7 open questions, and its information allows the estimation of the time spent per week in different dimensions of physical activity (walking and physical efforts of moderate and vigorous intensity) and physical inactivity (sitting position).
Mental health | From enrollment to the end of treatment at 6 weeks.
  The Mini Mental State Examination (MMSE) is a screening instrument to assess the domains (spatial and temporal orientation, immediate and recall memory, calculation, language-naming, repetition, comprehension, writing, and copying of drawings). The MMSE is a cognitive screening test that assesses cognitive function and may indicate dementia. The total score ranges from 0 to 30, with scores above 25 indicating normal cognitive function. Score Interpretation: 26-30 points: Normal cognitive function. 21-24 points: Mild cognitive impairment. 10-20 points: Moderate cognitive impairment. Less than or equal to 9 points: Severe cognitive impairment. Low or very low scores: Strong correlation with dementia, but other mental disorders may also affect the result.
Anterior Trunk Flexion Test | From enrollment to the end of treatment at 6 weeks.
  The Anterior trunk flexion test measures the distance between the tip of the middle finger and the floor after the participant performs forward trunk flexion with feet together and knees straight. The result is recorded in centimeters (cm) and uses the distance between the third finger and the floor. Unit of Measure: Centimeters (cm).
The Borg scale | From enrollment to the end of treatment at 6 weeks.
  The Borg scale is a numerical scale from "0" to "10", where the patient will indicate a score for their level of tiredness, at the beginning and end of each session, with "0" being no tiredness and "10" being maximum tiredness.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratório de Vibrações Mecânicas e Práticas Integrativas - LAVIMPI, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD supporting the results in publications will be utilized.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Available indefinitely.
Access Criteria: Unending.